CLINICAL TRIAL: NCT06595628
Title: Comparative Study of Modified Guarnieri-Desarda Technique Versus Lichtenstein Technique in Inguinal Hernia Repair
Brief Title: Modified Guarnieri-Desarda Technique Versus Lichtenstein Technique in Inguinal Hernia Repair
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Fadi Fawzi Azmi Khalil, Residend of Surgery, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MD-255-2022
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Inguinal Hernia
Keywords: Inguinal Hernia; Hernia Repair; Guarnieri Technique; Desarda Technique; Lichtenstein Hernioplasty
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Intervention Model Description: This study follows a parallel assignment model. Patients are randomly assigned to one of two groups: the Lichtenstein mesh-based repair group (L group) or the combined modified Guarnieri-Desarda tissue-based repair group (C group). The interventions are performed independently in each group, with outcomes compared between the two. There is no blinding in this study, and both the participants and the surgeons know which procedure is being performed (open-label study). The primary focus is on comparing the effectiveness and safety of the two surgical techniques.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lichtenstein Mesh-Based Repair (Active Comparator): Participants in this arm will undergo the Lichtenstein tension-free hernioplasty, which involves reinforcing the inguinal canal floor using a synthetic mesh. The mesh is fixed to the inguinal ligament and internal oblique aponeurosis, minimizing tension in the repair and reducing the risk of recurrence.
  Interventions: Procedure: Lichtenstein Mesh-Based Hernioplasty
- Combined Modified Guarnieri-Desarda Tissue-Based Repair (Experimental): Participants in this arm will receive the combined modified Guarnieri-Desarda tissue-based repair. This approach involves reconstructing the inguinal canal without the use of synthetic mesh, using the patient's own tissues to reinforce the canal and reduce tension. The technique combines aspects of both the Guarnieri and Desarda methods, aiming to preserve the natural physiology of the inguinal canal while providing tension-free repair.
  Interventions: Procedure: Combined Modified Guarnieri-Desarda Tissue-Based Hernioplasty

INTERVENTIONS:
Procedure: Lichtenstein Mesh-Based Hernioplasty — This is a tension-free hernioplasty procedure that uses a synthetic mesh to reinforce the inguinal canal floor. The mesh is fixed to the inguinal ligament and internal oblique aponeurosis, creating a barrier to prevent hernia recurrence. It is considered the gold standard for inguinal hernia repair and is widely used for its effectiveness in reducing recurrence rates and postoperative complications.
  Arms: Lichtenstein Mesh-Based Repair
Procedure: Combined Modified Guarnieri-Desarda Tissue-Based Hernioplasty — This technique combines elements of the Guarnieri and Desarda tissue-based repairs. It does not involve the use of synthetic mesh, relying instead on the patient's own tissues to reinforce the inguinal canal. The Guarnieri technique reshapes the internal ring to improve the inguinal canal's shutter mechanism, while the Desarda technique reinforces the posterior wall using the external oblique aponeurosis. This approach aims to preserve natural anatomy and minimize complications associated with mesh use.
  Arms: Combined Modified Guarnieri-Desarda Tissue-Based Repair

SUMMARY:
The aim of this study is to compare the surgical outcome of both Lichnichtien tension free mesh hernioplasty of inguinal hernia and the combined modified Guarnieri Desarda technique in terms of postoperative pain, post operative complications (seroma, hematoma, wound infection), chronic inguinodenia, early recurrence and assessment of testicular vascularity and size by application of a testicular duplex and ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Adult male patients aged 18 years or older.
* Patients diagnosed with non-complicated inguinal hernia (both direct and indirect).
* Patients able to provide written informed consent to participate in the study.

Exclusion Criteria:

* Patients younger than 18 years old.
* Patients with complicated hernias (e.g., inflamed, obstructed, or strangulated hernias).
* Patients with a recurrent inguinal hernia.
* Patients with weak or thin external oblique aponeurosis (intraoperative findings).
* Patients with a history of prior surgery in the inguinal region.
* Patients who refuse to participate in the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only individuals who self-identify as male are eligible to participate.
Enrollment: 40 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain Assessment | At 2 weeks, 1 month, 3 months, and 6 months post-surgery.
  Postoperative pain will be evaluated using the Mankoski Pain Scale (0-10). Pain scores will be recorded at different time intervals to assess immediate and long-term postoperative pain, with scores from 0 to 2 considered negligible, and scores from 3 to 10 considered significant.

SECONDARY OUTCOMES:
Incidence of Postoperative Complications | At 2 weeks, 1 month, and 3 months post-surgery.
  The occurrence of postoperative complications such as seroma, hematoma, wound infection, and testicular complications (e.g., hydrocele, cord induration) will be recorded and analyzed for each group.
Hernia Recurrence Rate | At 6 months and 1 year post-surgery.
  The rate of hernia recurrence will be assessed through clinical examination and imaging, comparing recurrence between the Lichtenstein mesh-based repair group and the modified Guarnieri-Desarda tissue-based repair group.
Testicular Vascularity | At 3 months post-surgery.
  Testicular vascularity will be evaluated using testicular duplex and ultrasound, comparing any changes pre- and post-surgery between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Fadi F. Khalil, MSc, Principal Investigator — Kasr El Aini Hospital
Locations (1):
- Kasralainy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) including demographic information, surgical outcomes, and follow-up data (postoperative pain scores, complications, testicular vascularity and size, and hernia recurrence rates) will be made available. Data will be shared with researchers upon reasonable request for the purpose of secondary analysis. Access to the data will be granted following the publication of the study results and will be available for up to 5 years after study completion. Participants' confidentiality will be protected, and any shared data will be anonymized.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available for a period of 5 years after the study is completed.
Access Criteria: Who: Qualified researchers with a scientifically sound proposal will be able to access the individual participant data (IPD) and supporting information.
  What: Researchers will be able to access de-identified IPD, including demographic data, surgical outcomes, follow-up data (e.g., pain scores, complications, testicular vascularity, and hernia recurrence), and supporting documents such as the study protocol, statistical analysis plan, and informed consent form.
  How: Researchers must submit a formal request to the corresponding author detailing their research proposal, the objectives of the secondary analysis, and how the data will be used. Requests will be evaluated by the study investigators. If approved, data will be shared via a secure, password-protected data-sharing platform, ensuring compliance with data protection regulations.